CLINICAL TRIAL: NCT00619476
Title: Study PXN110748: An Efficacy and Safety Study of XP13512 Compared With a Concurrent Placebo Control in Subjects With Neuropathic Pain Associated With Post-herpetic Neuralgia (PHN)
Brief Title: A Study In Patients With Neuropathic Pain From Post-Herpetic Neuralgia (PHN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 110748
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Results first posted 2011-05-20 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-01

CONDITIONS: Neuralgia, Postherpetic
Keywords: Neuropathic Pain; Post-herpetic neuralgia; PHN
MeSH Terms: conditions — Neuralgia, Postherpetic; Neuralgia | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo
- GEn 1200mg/day (Experimental): gabapentin enacarbil 1200mg/day, maintenance treatment 14 weeks
  Interventions: Drug: GEn 1200mg/day
- GEn 2400mg/day (Experimental): gabapentin enacarbil 2400mg/day, maintenance treatment 14 weeks
  Interventions: Drug: GEn 2400mg/day
- GEn 3600mg/day (Experimental): gabapentin enacarbil 3600mg/day, maintenance treatment 14 weeks
  Interventions: Drug: GEn 3600mg/day

INTERVENTIONS:
Drug: GEn 1200mg/day — gabapentin enacarbil 1200mg/day
  Other Names: XP13512/GSK1838262; gabapentin enacarbil
  Arms: GEn 1200mg/day
Drug: GEn 2400mg/day — gabapentin enacarbil 2400mg/day
  Other Names: XP13512/GSK1838262; gabapentin enacarbil
  Arms: GEn 2400mg/day
Drug: GEn 3600mg/day — gabapentin enacarbil 3600mg/day
  Other Names: gabapentin enacarbil; XP13512/GSK1838262
  Arms: GEn 3600mg/day
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether gabapentin enacarbil (XP13512/GSK1838262), hereafter referred to as GEn is effective in the treatment of neuropathic pain associated with post-herpetic neuralgia (PHN).

DETAILED DESCRIPTION:
The primary purpose of study PXN110748 was to evaluate efficacy and safety of 3 fixed doses of GEn in the treatment of PHN.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Female subjects are eligible if of non-childbearing potential or not lactating, has a negative pregnancy, and agrees to use one a specified highly effective method for avoiding pregnancy
* Documented medical diagnosis of PHN of with pain present for at least three months from the healing of a herpes zoster rash
* Baseline 24-hour average pain intensity score ≥ 4.0 based on an 11-point PI-NRS
* Provides written informed consent in accordance with all applicable regulatory requirements

Exclusion Criteria:

* Other chronic pain conditions not associated with PHN. However, the subject will not be excluded if:
* The pain is located at a different region of the body; and
* The pain intensity is not greater than the pain intensity of the PHN; and
* The subject can assess PHN pain independently of other pain
* Is unable to discontinue prohibited medications or non-drug therapies or procedures throughout the duration of the study
* Hepatic impairment defined as ALT or AST > 2x upper limit of normal (ULN), or alkaline phosphatase or bilirubin > 1.5x ULN
* Chronic hepatitis B or C
* Impaired renal function defined as creatinine clearance <60 mL/min or requiring hemodialysis
* Corrected QT (QTc) interval ≥ 450 msec or QTc interval ≥480 msec for patients with Bundle Branch Block
* Uncontrolled hypertension at screen (sitting systolic >160 mmHg and/or sitting diastolic >90 mmHg)
* Current diagnosis of active epilepsy or any active seizure disorder requiring chronic therapy with antiepileptic drugs
* Medical condition or disorder that would interfere with the action, absorption, distribution, metabolism, or excretion of GEn, or, in the investigator's judgment
* Is considered to be clinically significant and may pose a safety concern, or,
* Could interfere with the accurate assessment of safety or efficacy, or,
* Could potentially affect a subject's safety or study outcome
* Meets criteria defined by the DSM-IV-TR for a major depressive episode or for active significant psychiatric disorders within last year
* Depression in remission, with or without antidepressant treatment, may participate, unless stable antidepressant regimen is a prohibited medication
* Antidepressant medication may not be changed or discontinued to meet entry criteria and must be stable for at least three months prior to enrollment
* History of clinically significant drug or alcohol abuse (DSM-IV-TR) or is unable to refrain from substance abuse throughout the study. Benzodiazepines or atypical benzodiazepines as hypnotic sleep agents permitted.
* Currently participating in another clinical study in which the subject is, or will be exposed to an investigational or non-investigational drug or device
* Has participated in a clinical study and was exposed to investigational or non-investigational drug or device:
* Within preceding month for studies unrelated to PHN, or
* Within preceding six months for studies related to PHN
* Treated previously with GEn
* History of allergic or medically significant adverse reaction to investigational products (including gabapentin) or their excipients, acetaminophen or related compounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2008-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (79):
- United States (68):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Northport, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Litchfield Park, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Arcadia, California
  - GSK Investigational Site, Huntington Park, California
  - GSK Investigational Site, New Port Beach, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Oxnard, California
  - GSK Investigational Site, Redondo Beach, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Boulder, Colorado
  - GSK Investigational Site, Bradenton, Florida
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Hallandale, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Naranja, Florida
  - GSK Investigational Site, New Port Richey, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Libertyville, Illinois
  - GSK Investigational Site, Danville, Indiana
  - GSK Investigational Site, Elkhart, Indiana
  - GSK Investigational Site, Terre Haute, Indiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Bingham Farms, Michigan
  - GSK Investigational Site, Olive Branch, Mississippi
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Reno, Nevada
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Amherst, New York
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, High Point, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Norman, Oklahoma
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Altoona, Pennsylvania
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Weber City, Virginia
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Wenatchee, Washington
  - GSK Investigational Site, Yakima, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
- Canada (11):
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Niagara Falls, Ontario
  - GSK Investigational Site, Thornhill, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint Romuald, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Three 600 milligram (mg) gabapentin enacarbil (XP13512/GSK1838262), hereafter referred to as GEn, placebo tablets taken orally twice daily (morning and evening)
- GEn 1200 mg/Day: One 600 mg GEn tablet and two GEn placebo tablets taken orally twice daily (morning and evening)
- GEn 2400 mg/Day: Two 600 mg GEn tablets and one GEN placebo tablet taken orally twice daily (morning and evening)
- GEn 3600 mg/Day: Three 600 mg GEn tablets taken orally twice daily (morning and evening)
Period: Overall Study
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Started | 95 | 107 | 84 | 90
Intent-to-Treat Population | 95 | 107 | 82 | 87
Safety Population | 95 | 107 | 82 | 87
Completed | 64 | 85 | 60 | 56
Not Completed | 31 | 22 | 24 | 34
Not completed — Adverse Event | 12 | 6 | 12 | 16
Not completed — Lack of Efficacy | 6 | 1 | 1 | 4
Not completed — Protocol Violation | 5 | 4 | 4 | 9
Not completed — Lost to Follow-up | 1 | 2 | 0 | 1
Not completed — Investigator Discretion | 2 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 5 | 7 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day | Total
Number analyzed (Participants) | 95 | 107 | 82 | 87 | 371
Age Continuous [Mean (Standard Deviation); unit: Years] — Age in years of the Intent-to-Treat (ITT) Population, comprised of all randomized participants who took at least one dose of investigational product and provided at least one post-baseline efficacy measurement, was used for all baseline characteristics.
  Years | 61.7 (12.77) | 61.7 (12.58) | 64.1 (8.94) | 61.3 (15.41) | 62.1 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender of the ITT Population, comprised of all randomized participants who took at least one dose of investigational product and provided at least one post-baseline efficacy measurement, was used for all baseline characteristics.
  Participants
    Female | 45 | 54 | 35 | 48 | 182
    Male | 50 | 53 | 47 | 39 | 189
Race/Ethnicity, Customized [Number; unit: participants] — Race of the ITT Population, comprised of all randomized participants who took at least one dose of investigational product and provided at least one post-baseline efficacy measurement, was used for all baseline characteristics.
  participants
    White | 79 | 94 | 69 | 73 | 315
    African American/African Heritage | 14 | 11 | 8 | 11 | 44
    American Indian or Alaskan Native | 0 | 0 | 2 | 1 | 3
    Asian - Central/South Asian Heritage | 1 | 0 | 1 | 0 | 2
    Asian - Japanese/ East Asian Heritage | 0 | 1 | 1 | 1 | 3
    Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 1 | 1
    Not Provided | 1 | 1 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Mean 24-hour Average Pain Intensity (API) Score at the End of Maintenance Treatment (EOMT) Using Last Observation Carried Forward (LOCF) Data
Description: Baseline and EOMT values are the calculated means of the daily 24-hour API scores for each participant during the last 7 days prior to randomization (Baseline) and the earliest date of Week 13 visit/Withdrawal visit/last dose of study drug (EOMT). Participants used a hand-held diary to rate their average pain intensity over the preceding 24 hours, using an 11-point PI-Numerical Rating Scale (0=no pain, 10=pain as bad as you can imagine). LOCF was used if less than 4 days of diary data were provided. Change from baseline was calculated as EOMT score minus Baseline score.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population: all randomized participants who took at least one dose of investigational product and provided at least one post-baseline efficacy measurement.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Number analyzed (Participants) | 95 | 107 | 82 | 87
points on a scale | -1.66 (0.216) | -2.47 (0.204) | -2.36 (0.237) | -2.72 (0.227)
Statistical Analysis 1: Comparison: Placebo vs GEn 1200 mg/Day; Test type: Superiority or Other; p = 0.013, ANCOVA — This p-value has been adjusted for multiplicity using a step-down procedure that uses Dunnett's test within a closed testing scheme for multiple comparisons with a common control in order to maintain the overall experiment-wise alpha level of 0.05; An ANCOVA model with body mass index (BMI), baseline 24-hour average pain intensity, and grouped center as covariates was used; Adjusted Mean difference versus placebo = -0.81, 95% CI 2-sided [-1.40 to -0.23]
Statistical Analysis 2: Comparison: Placebo vs GEn 2400 mg/Day; Test type: Superiority or Other; p = 0.029, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted Mean difference versus placebo = -0.70, 95% CI 2-sided [-1.33 to -0.07]
Statistical Analysis 3: Comparison: Placebo vs GEn 3600 mg/Day; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Adjusted Mean difference versus placebo = -1.07, 95% CI 2-sided [-1.68 to -0.45]

2. Secondary Outcome: Change From Baseline in the Mean Night-time Average Pain Intensity (API) Score at EOMT Using LOCF Data
Description: Night-time is defined as the time between going to bed at night and rising in the morning. Participants recorded night-time API on a daily basis in the morning upon awakening using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Baseline and EOMT are as defined for the primary endpoint. Change from baseline wss calculated as the EOMT score minus the baseline score. An ANCOVA model with baseline value, BMI, grouped center as covariates was used.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. There was one participant in the GEn 2400 mg group and one in the 3600 mg group who did not complete enough post-baseline morning diaries to calculate an API for the EOMT timepoint.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Number analyzed (Participants) | 95 | 107 | 81 | 86
points on a scale | -1.65 (0.219) | -2.35 (0.206) | -2.44 (0.238) | -2.50 (0.231)

3. Secondary Outcome: Change From Baseline in the Mean Current Morning Pain Intensity Score at EOMT Using LOCF Data
Description: Current pain is defined as the participant's assessment of pain intensity "right now." Participants recorded their current morning pain intensity in the morning upon wakening using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Baseline and EOMT are as defined for the primary endpoint. Change from baseline was calculated as the EOMT score minus the baseline score. An ANCOVA model with baseline value, BMI, grouped center as covariates was used.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. There was one participant in the GEn 2400 mg group and one in the 3600 mg group who did not complete enough post-baseline morning diaries to calculate an API for the EMOT timepoint.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Number analyzed (Participants) | 95 | 107 | 81 | 86
points on a scale | -1.34 (0.223) | -2.29 (0.209) | -2.13 (0.242) | -2.41 (0.234)

4. Secondary Outcome: Change From Baseline in the Mean Night-time Worst Pain Intensity Score at EOMT Using LOCF Data
Description: Night-time worst pain is defined as the participant's assessment of their worst pain between going to bed at night and rising in the morning. Participants recorded night-time worst pain in the morning upon awakening using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Baseline and EOMT are as defined for the primary endpoint. Change from baseline was calculated as the EOMT score minus the baseline score. An ANCOVA model with baseline value, BMI, grouped center as covariates was used.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Number analyzed (Participants) | 95 | 107 | 81 | 86
points on a scale | -1.76 (0.239) | -2.49 (0.225) | -2.65 (0.260) | -2.71 (0.252)

5. Secondary Outcome: Change From Baseline in the Mean Sleep Interference Score at EOMT Using LOCF Data
Description: Participants assessed sleep interference due to pain on a daily basis using the 11-point NRS (0=pain does not interfere with sleep, 10=pain completely interferes with sleep). Baseline and EOMT are as defined for the primary endpoint. Change from baseline was calculated as the EOMT score minus the baseline score. An ANCOVA model with baseline value, BMI, grouped center as covariates was used.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. There was one participant in the GEn 2400 mg group and one in the 3600 mg group who did not complete enough post-baseline morning diaries to calculate a score for the EMOT timepoint.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Number analyzed (Participants) | 95 | 107 | 81 | 86
points on a scale | -2.04 (0.225) | -2.72 (0.212) | -2.58 (0.245) | -2.78 (0.237)

6. Secondary Outcome: Change From Baseline in the Mean Day-time Average Pain Intensity(API) Score at EOMT Using LOCF Data
Description: Day-time is defined as the time between rising in the morning and going to bed at night. Participants recorded day-time API on a daily basis in the evening before bedtime using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Baseline and EOMT are as defined for the primary endpoint. Change from baseline was calculated as the EOMT score minus the baseline score. An ANCOVA model with baseline value, BMI, grouped center as covariates was used.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. There was one participant in the GEn 1200 mg group and two in the 2400 mg group who did not complete enough post-baseline evening diaries to calculate an API for the EOMT timepoint.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Number analyzed (Participants) | 95 | 106 | 80 | 87
points on a scale | -1.59 (0.218) | -2.47 (0.206) | -2.23 (0.239) | -2.67 (0.229)

7. Secondary Outcome: Change From Baseline in the Mean Current Evening Pain Intensity Score at EOMT Using LOCF Data
Description: Current pain is defined as the participant's assessment of pain intensity "right now." Participants recorded their current evening pain intensity in the evening before bedtime using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Baseline and EOMT are as defined for the primary endpoint. Change from baseline was calculated as the EOMT score minus the baseline score. An ANCOVA model with baseline value, BMI, grouped center as covariates was used.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. There was one participant in the GEn 1200 mg group and two in the 2400 mg group who did not complete enough post-baseline evening diaries to calculate a score for the EMOT timepoint.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Number analyzed (Participants) | 95 | 106 | 80 | 87
points on a scale | -1.45 (0.225) | -2.45 (0.213) | -2.24 (0.247) | -2.69 (0.236)

8. Secondary Outcome: Change From Baseline in the Mean Day-time Worst Pain Intensity Score at EOMT Using LOCF Data
Description: Day-time worst pain is defined as the participant's assessment of their worst pain between rising in the morning and going to bed at night. Participants recorded day-time worst pain in the evening before bedtime using an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Baseline and EOMT are as defined for the primary endpoint. Change from baseline was calculated as the EOMT score minus the baseline score. An ANCOVA model with baseline value, BMI, grouped center as covariates was used.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. There was one participant in the GEn 1220 mg group and two in the 2400 mg group who did not complete enough post-baseline evening diaries to calculate a score for the EOMT timepoint.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Number analyzed (Participants) | 95 | 106 | 80 | 87
points on a scale | -1.74 (0.242) | -2.61 (0.229) | -2.41 (0.265) | -2.82 (0.253)

9. Secondary Outcome: Change From Baseline in Pain Quality as Assessed by the Neuropathic Pain Scale (NPS) Summary Scores at EOMT Using LOCF Data
Description: The NPS assesses pain qualities and consists of 11-items, 10 assessed on an 11-point NRS (0=no impact to 10=greatest impact); and 1 open-ended question not used in score calculation. 4 summary scores are calculated: NPS 10 (items 1-7, 9-11), NPS 8 (8 pain descriptor items), NPS Non-Allodynic (NA) (8 NA items), and NPS 4 (4 pain quality items); and range from 0 to 100 (0=no impact and 100=greatest impact). The analysis is based on the change from baseline (BL) (EOMT score minus the BL score) using an ANCOVA model with BL value, BMI, grouped center as covariates.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. The NPS summary included a subset of the ITT Population that completed an NPS assessment at both Baseline and Week 13/Withdrawal.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Number analyzed (Participants) | 85 | 102 | 74 | 77
points on a scale
  NPS 10 Score | -17.17 (2.094) | -22.78 (1.907) | -24.02 (2.256) | -25.2 (2.202)
  NPS 8 Score | -17.05 (2.059) | -22.23 (1.875) | -23.77 (2.217) | -24.49 (2.165)
  NPS Non-Allodynic Score | -16.87 (2.107) | -22.58 (1.920) | -24.18 (2.269) | -24.54 (2.216)
  NPS 4 Score | -18.25 (2.340) | -24.37 (2.133) | -26.08 (2.519) | -26.55 (2.464)

10. Secondary Outcome: Change From Baseline in Pain Characteristics and Intensity as Assessed by the Short Form-McGill Pain Questionnaire (SF-MPQ) at EOMT Using LOCF Data
Description: The SF-MPQ, a general pain instrument, assesses the characteristics and intensity of pain and consists of 15-items assessed on a 4-point scale (0=none, 1=mild, 2=moderate, and 3=severe). 3 summary scores are calculated: sensory score (sum of items 1-11, range 0-33), affective score (sum of items 12-15, range 0-12), total score (sum of items 1-15, range 0-45), where lower scores = lower pain/impact. Analysis is based on the change from baseline (BL) (EOMT score minus the BL score) using an ANCOVA model with BL value, BMI, grouped center as covariates.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. The SF-MPQ analysis included a subset of the ITT Population who completed a SF-MPQ assessment at both Baseline and the Week 13/Withdrawal Visit.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Number analyzed (Participants) | 85 | 101 | 74 | 76
points on a scale
  SF-MPQ Total Score | -6.08 (0.949) | -8.35 (0.869) | -7.45 (1.024) | -8.15 (1.006)
  SF-MPQ Sensory Score | -4.51 (0.737) | -6.07 (0.675) | -5.43 (0.795) | -6.13 (0.782)
  SF-MPQ Affective Score | -1.58 (0.270) | -2.27 (0.247) | -2.08 (0.291) | -1.99 (0.286)

11. Secondary Outcome: Change From Baseline in Dynamic Allodynia at EOMT Using LOCF Data
Description: Dynamic allodynia (pain in response to a standardized light touch stimulus, a foam brush applied with light pressure to the site of maximum pain) was assessed by an 11-point PI-NRS (0=no pain, 10=pain as bad as you can imagine). Baseline and EOMT are as defined for the primary endpoint. Change from baseline was calculated as the EOMT score minus the baseline score. An ANCOVA model with baseline value, BMI, grouped center as covariates was used.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. The NRS analysis included a subset of the ITT Population who completed that NRS at both the Baseline and the Week13/Withdrawal Visit.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Number analyzed (Participants) | 85 | 100 | 73 | 74
points on a scale | -2.29 (0.150) | -1.97 (0.137) | -2.16 (0.161) | -2.25 (0.161)

12. Secondary Outcome: Number of Participants Who Are Responders on the Patient Global Impression of Change (PGIC) Questionnaire at EOMT Using LOCF Data
Description: The PGIC is a single-item questionnaire designed to provide an overall assessment of treatment from the participant's perspective since the start of the study. It is measured on a 7-point scale, where 1=very much improved and 7=very much worse. A participant is considered a responder if they have a response of "very much improved" or "much improved." EOMT response is defined as the score recorded at the Week13/Withdrawal visit.
Time Frame: EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. The PGIC analysis included a subset of the ITT Population who completed the PGIC questionnaire at the end of treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Number analyzed (Participants) | 85 | 103 | 78 | 76
participants | 24 | 45 | 35 | 39

13. Secondary Outcome: Number of Participants Achieving Various Levels of Percent Reduction From Baseline in the Mean 24-hour Average Pain Intensity Score at EOMT Using LOCF Data
Description: Baseline and EOMT scores are the calculated means of the 24-hour average pain scores for each participant during the last 7 days prior to randomization and EOMT, respectively. Percent reduction from baseline was calculated as the [(EOMT score minus the baseline score)divided by the baseline score], multiplied by 100. The PI-NRS is an 11-point scale (0=no pain, 10=pain as bad as you can imagine) by which a participant assesses their 24-hour average pain intensity.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. There was one participant in the GEn 1200 mg and one in the GEn 2400 mg group who did not have enough data available to calculate the percent reduction.
Measure: Number; unit: participants
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Number analyzed (Participants) | 95 | 106 | 81 | 87
participants
  >=0 reducation from baseline | 79 | 94 | 71 | 84
  >= 10% reduction from baseline | 62 | 83 | 61 | 70
  >= 20% reduction from baseline | 50 | 71 | 55 | 65
  >= 30% reduction from baseline | 40 | 57 | 48 | 52
  >= 40% reduction from baseline | 32 | 50 | 39 | 46
  >= 50% reduction from baseline | 22 | 44 | 28 | 37
  >= 60% reduction from baseline | 15 | 34 | 14 | 31
  >= 70% reduction from baseline | 9 | 25 | 18 | 24
  >= 80% reduction from baseline | 8 | 17 | 12 | 19
  >= 90% reduction from baseline | 3 | 9 | 9 | 12
  100% reduction from baseline | 1 | 6 | 3 | 7

14. Secondary Outcome: Time to Onset of Sustained Improvement in the 24-hour Average Pain Intensity Score
Description: Sustained improvement in the 24-hour average pain intensity score is defined as at least 2 consecutive days on which the 24-hour average pain intensity score is >=2 points less than the mean 24-hour average pain intensity score at baseline. Time to onset is measured from baseline and was calculated as the first day of event minus the last day of baseline and is expressed in days. Baseline score is the calculated mean of the 24-hour average pain score for each participant during the last 7 days prior to randomization.
Time Frame: Anytime post-baseline until date of last dose of study medication (up to Week 13)
Population: ITT Population
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Number analyzed (Participants) | 95 | 107 | 82 | 87
days | 49 [2 to 86] | 27 [1 to 96] | 10 [1 to 79] | 10 [1 to 67]

15. Secondary Outcome: Change From Baseline in the Mean Daily Dose in Milligrams of Rescue Medication at EOMT Using LOCF Data
Description: Mean daily use of rescue medication (milligrams of acetaminophen) was calculated by determining the average number of tablets taken per day of rescue medication (Commerical Tylenol) during treatment and multiplying that by 500 mg. Baseline and EOMT are as defined for the primary endpoint. Change from baseline was calculated as the EOMT score minus the baseline score. An ANCOVA model with baseline value, BMI, grouped center as covariates was used.
Time Frame: Baseline and EOMT (Week 13 or early withdrawal)
Population: ITT Population. There was one participant in the GEn 1200 mg and two in the GEn 2400 mg group who did not have enough data available to calculate the rescue mediation consumed while on treatment.
Measure: Least Squares Mean (Standard Error); unit: milligrams
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Number analyzed (Participants) | 95 | 106 | 80 | 87
milligrams | -41.00 (89.488) | -289.94 (84.350) | -260.03 (97.853) | -266.21 (93.503)

16. Secondary Outcome: Change From Baseline in Severity of Pain and the Impact of Pain as Assessed by the Brief Pain Inventory (BPI) at EOMT Using LOCF Data
Description: The BPI, a general pain instrument, assesses the severity and interference of pain; and consists of 6 items assessed on an 11-point NRS (0=no impact and 10=greatest impact). 2 summary scores are calculated: BPI Severity Score (average of first 4 items) and BPI Interference Score (average of 7 responses to item 6); where each summary score ranges from 0 to 10 (0=no impact and 10=greatest impact). Analysis of this endpoint is based on the change from baseline (BL) (EOMT score minus the BL score) using an ANCOVA model with BL value, BMI, grouped center as covariates.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. Not all participants completed a BPI assessment at both Baseline and Week 13/Withdrawal; as such, the number analyzed is different from the full ITT Population counts.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Number analyzed (Participants) | 85 | 101 | 74 | 76
points on a scale
  Brief Pain Inventory Severity of Pain | -1.8 (0.22) | -2.4 (0.20) | -2.4 (0.24) | -2.5 (0.24)
  Brief Pain Inventory Interference of Pain | -2.0 (0.20) | -2.2 (0.19) | -2.2 (0.22) | -2.3 (0.22)

17. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by the SF-36 at EOMT Using LOCF Data
Description: The SF-36 is a general health-related quality of life instrument consisting of 36 items with various response options (Yes/No, 5- to 6-point Likert scale). Summary scores are calculated for 8 domains and 2 components (physical and mental); where scores range from 0 to 100 (higher scores = better quality of life). Analysis of this endpoint is based on the change from baseline (BL) (EOMT score minus the BL score) using an ANCOVA model with BL value, BMI, grouped center as covariates.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. Not all participants completed an SF-36 at both Baseline and Week 13/Withdrawal; as such, the number analyzed is different from the full ITT Population counts.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Number analyzed (Participants) | 85 | 101 | 74 | 75
points on a scale
  SF-36 Physical Component Summary Score | 3.3 (0.74) | 4.3 (0.67) | 4.4 (0.79) | 4.9 (0.78)
  SF-36 Mental Component Summary Score | 3.2 (0.92) | 5.1 (0.85) | 4.5 (0.99) | 5.8 (0.99)

18. Secondary Outcome: Change From Baseline in Emotional Functioning as Assessed by the POMS-B at EOMT Using LOCF Data
Description: The POMS-B, an emotional functioning instrument, assesses mood, tension, and other psychological symptoms and consists of 30-items assessed on a 5-point scale (0=not at all to 4=extremely). 6 summary scores are calculated: Tension/Anxiety, Depression/Rejection, Anger/Hostility, Vigor/Activity, Fatigue/Inertia, and Confusion/Bewilderment; and range from 0-20 (higher scores = more negative mood state). Analysis of this endpoint is based on the change from baseline (BL) (EOMT score minus the BL score) using an ANCOVA model with BL value, BMI, grouped center as covariates.
Time Frame: Baseline and EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. Not all participants completed a POMS-B at both Baseline and Week 13/Withdrawal; as such, the number analyzed is different from the full ITT Population counts.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Number analyzed (Participants) | 85 | 101 | 74 | 75
points on a scale
  Tension/Anxiety Domain Score | -1.6 (0.29) | -1.8 (0.26) | -2.0 (0.30) | -2.0 (0.30)
  Depression/Rejection Domain Score | -1.4 (0.28) | -1.5 (0.26) | -1.9 (0.30) | -1.7 (0.30)
  Anger/Hostility Domain Score | -1.6 (0.29) | -2.0 (0.27) | -2.4 (0.31) | -1.7 (0.31)
  Vigor/Activity Domain Score | 0.4 (0.38) | 0.8 (0.35) | 0.5 (0.41) | 1.4 (0.41)
  Fatigue/Inertia Domain Score | -1.4 (0.40) | -1.9 (0.37) | -2.4 (0.43) | -2.5 (0.43)
  Confusion/Bewilderment Domain Score | -0.7 (0.25) | -0.5 (0.22) | -1.0 (0.26) | -0.5 (0.26)

19. Secondary Outcome: Number of Participants Who Are Responders on the Clinician Global Impression of Change (CGIC) Questionnaire at EOMT Using LOCF Data
Description: The CGIC is a single-item questionnaire designed to provide an overall assessment of treatment from the clinician's perspective since the start of the study. It is measured on a 7-point scale, where 1=very much improved and 7=very much worse. A participant is considered a responder if they have a response of "very much improved" or "much improved." EOMT response is defined as the score recorded at the Week13/Withdrawal visit.
Time Frame: EOMT (representing the earliest date of Week 13 visit/withdrawal visit)
Population: ITT Population. The CGIC analysis included a subset of the ITT Population who completed the PGIC questionnaire at the end of treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Number analyzed (Participants) | 68 | 85 | 68 | 68
participants | 21 | 38 | 34 | 33

ADVERSE EVENTS:
Description: Adverse Events (AEs) and serious adverse events (SAEs) were captured for all participants in the Safety Population, which was comprised of all randomized participants who took at least one dose of investigational product.
Arm/Group | Placebo | GEn 1200 mg/Day | GEn 2400 mg/Day | GEn 3600 mg/Day
Serious Adverse Events (participants affected / at risk) | 2/95 | 0/107 | 6/82 | 2/87
Other Adverse Events (participants affected / at risk) | 63/120 | 75/107 | 64/82 | 71/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=95) | GEn 1200 mg/Day (N=107) | GEn 2400 mg/Day (N=82) | GEn 3600 mg/Day (N=87)
Intracranial Aneruysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 | 0 (0)
Multiple Sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 | 0 (0)
Vascular Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 (0) | 0 (0)
Blood Pressure Increased (Investigations) | 0 (0) | 0 (0) | 1 | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=120) | GEn 1200 mg/Day (N=107) | GEn 2400 mg/Day (N=82) | GEn 3600 mg/Day (N=87)
Dizziness (Nervous system disorders) | 14 | 18 | 21 | 26
Somnolence (Nervous system disorders) | 8 | 11 | 9 | 12
Headache (Nervous system disorders) | 9 | 11 | 8 | 6
Nausea (Gastrointestinal disorders) | 5 | 9 | 3 | 8
Constipation (Gastrointestinal disorders) | 5 | 7 | 4 | 4
Diarrhea (Gastrointestinal disorders) | 5 | 6 | 2 | 6
Fatigue (General disorders) | 1 | 5 | 4 | 9
Nasopharyngitis (Infections and infestations) | 5 | 5 | 3 | 5
Edema Peripheral (General disorders) | 0 (0) | 6 | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 6 | 4 | 3
Insomnia (Psychiatric disorders) | 2 | 3 | 4 | 6
Urinary Tract Infection (Infections and infestations) | 3 | 8 | 2 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 4 | 2
Weight Increased (Investigations) | 1 | 3 | 4 | 4
Dry Mouth (Gastrointestinal disorders) | 2 | 1 | 4 | 4
Hypertension (Cardiac disorders) | 1 | 2 | 4 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 5
Vision Blurred (Eye disorders) | 0 (0) | 2 | 4 | 2
Flatulance (Gastrointestinal disorders) | 0 (0) | 1 | 1 | 4
Joint Sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 | 0 (0) | 4
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.